CLINICAL TRIAL: NCT06550895
Title: A Phase 2, Open-Label, Multicenter Study of Ciltacabtagene Autoleucel and Talquetamab for the Treatment of Participants With High-Risk Multiple Myeloma
Brief Title: A Study of Ciltacabtagene Autoleucel and Talquetamab for the Treatment of Participants With High-Risk Multiple Myeloma
Acronym: MonumenTAL-8
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 64407564MMY2008; 64407564MMY2008 (Other: Janssen Research & Development, LLC); 2023-507989-76-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1:Cilta-cel + Talquetamab Consolidation Post Chimeric Antigen Receptor T cell (CAR-T) Therapy (Experimental): Participants with relapsed and/or refractory multiple myeloma (RRMM) will be administered Cilta-cel followed by multiple cycles of talquetamab consolidation treatment and will be followed up until death, lost to follow-up, consent withdrawal, or study end, whichever occurs first.
  Interventions: Drug: Cilta-cel; Drug: Talquetamab

INTERVENTIONS:
Drug: Cilta-cel — Cilta-cel infusion will be administered intravenously.
  Other Names: Ciltacabtagene autoleucel, JNJ-68284528
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
  Other Names: JNJ-64407564

SUMMARY:
The purpose of this study is to define the safety of Ciltacabtagene Autoleucel (Cilta-cel) and Talquetamab in participants with high-risk multiple myeloma (MM).

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of MM according to the IMWG diagnostic criteria and is defined as a measurable disease at screening
* Cohort 1: Received at least 3 prior lines of antimyeloma therapy and have undergone greater than or equal to (>=) 1 complete cycle of the therapy
* Cohort 1: Documented evidence of progression of disease (PD) or failure to achieve a response to the last line of therapy
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Participant of childbearing potential (POCBP) must have a negative pregnancy test using a highly sensitive β-human chorionic gonadotropin (hCG) serum pregnancy test at screening

Exclusion Criteria:

* Cohort 1: Prior treatment with chimeric antigen receptor T cell (CAR-T) therapy directed at any target or any prior B cell maturation antigen (BCMA)-directed therapy/prior G protein-coupled receptor family C Group 5 member D (GPRC5D)-directed therapy
* Cohort 1: Received either of the following: An allogenic stem cell transplant within 6 months before apheresis/first dose of study drug and no immunosuppressive medications administered before the start of study treatment. And secondly, received an autologous stem cell transplant less than (<)12 weeks before apheresis/first dose of study treatment
* Receive live, attenuated vaccine within 4 weeks of enrollment
* Toxicity from previous anticancer therapy not resolved to baseline levels or to Grade 1 or less except for alopecia or peripheral neuropathy
* Stroke, transient ischemic attack, or seizure within 6 months of signing informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AE) by Severity According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 | Up to 3 years and 5 months
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical (investigational or non-investigational) product. It does not necessarily have a causal relationship with the investigational product. The severity of AEs has 5 grades based on NCI-CTCAE version 5.0 criteria: Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4: Life-threatening consequences; Grade 5: Death.

SECONDARY OUTCOMES:
Percentage of Participants With Overall Response (OR) | Up to 3 years and 5 months
  The percentage of participants who have a partial response (PR) or better response according to the International Myeloma Working Group (IMWG) response criteria will be reported.
Percentage of Participants with Very Good Partial Response (VGPR) or Better | Up to 3 years and 5 months
  The percentage of participants who achieve a VGPR or better response according to the IMWG response criteria will be reported.
Percentage of Participants with Complete Response (CR) or Stringent Complete Response (sCR) | Up to 3 years and 5 months
  The percentage of participants with best overall response of CR or sCR will be reported according to IMWG criteria.
Duration of Response (DOR) | Up to 3 years and 5 months
  DOR is defined as the time from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease (PD) (defined in the IMWG response criteria) or death due to any cause, whichever occur first.
Time to Response (TTR) | Upto 3 years and 5 months
  TTR is defined as the time between date of the first study treatment and the first efficacy evaluation that the participant met all criteria for PR or better.
Progression Free Survival (PFS) | Up to 3 years and 5 months
  PFS is defined as the time from the date of the first study treatment to the date of first documented disease progression (defined in the IMWG response criteria), or death due to any cause, whichever occurs first.
Overall Survival | Up to 3 years and 5 months
  Overall Survival is measured from the date of the first study treatment to the date of the participant's death.
Percentage of Participants with Minimal Residual Disease (MRD) Negativity | Up to 3 years and 5 months
  The percentage of participants who achieve MRD-negativity at a threshold of 10^-5 at any timepoint after the date of the first study treatment and before disease progression or start of any subsequent antimyeloma therapy will be reported.
Percentage of Participants with Sustained MRD-Negativity | Up to 3 years and 5 months
  The percentage of participants who sustained MRD-negative status, as determined by next generation sequencing (NGS) with sensitivity of 10^-5, for at least 6 months without examination showing MRD-positive or PD in between will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- United States (5):
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Australia (4):
  - Royal Prince Alfred Hospital, Camperdown
  - Austin Hospital, Heidelberg
  - Peter MacCallum Cancer Centre, Melbourne
  - The Alfred Hospital, Melbourne

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency